CLINICAL TRIAL: NCT02626871
Title: Atrial Fibrillation, Stroke, and Bleeding in Patients Undergoing Aortic Biovalve Implantation
Acronym: CAREAVR
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Helsinki University Central Hospital (Other); Oulu University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Tuomas Kiviniemi, MD, PhD, University of Turku
Other Study IDs: T39/2015
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation; Stroke; Transient Ischemic Attack; Bleeding; Aortic Stenosis
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Attack, Transient; Hemorrhage; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of the FIN-bioAVR registry is to assess the incidence of AF, strokes and major bleeding events in patients undergoing aortic valve replacement. This retrospective multicenter registry will include 850 patients with aortic valve replacement using bioprosthesis.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing aortic valve bioprosthesis implantation

Exclusion Criteria:

* mechanical heart valves in any position

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers design of patients undergoing aortic valve bioprosthesis implantation
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2002-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Stroke | 10 years
Mortality | 10 years
atrial fibrillation | 10 years
major bleeding | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Kiviniemi, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bjorn R, Lehto J, Malmberg M, Anttila V, Airaksinen KEJ, Gunn J, Kiviniemi T. Antithrombotic Medication and Major Complications After Mechanical Aortic Valve Replacement. Am J Cardiol. 2023 Oct 1;204:185-194. doi: 10.1016/j.amjcard.2023.07.097. Epub 2023 Aug 4. PMID 37544143
- [Derived] Salmi SJ, Nieminen T, Hartikainen J, Biancari F, Lehto J, Nissinen M, Malmberg M, Yannopoulos F, Savolainen J, Airaksinen J, Kiviniemi T. Indications and predictors for pacemaker implantation after isolated aortic valve replacement with bioprostheses: the CAREAVR study. Interact Cardiovasc Thorac Surg. 2020 Sep 1;31(3):398-404. doi: 10.1093/icvts/ivaa119. PMID 32747953